CLINICAL TRIAL: NCT04393324
Title: The Critical Care Resources Adaptation to the SARS-CoV-2 Pandemic in Madrid
Brief Title: The Critical Care Response to the COVID-19 Pandemic in Madrid
Acronym: Tetrix
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: FUNDACION PARA LA INVESTIGACION HOSPITAL CLINICO SAN CARLOS (Other)
Responsible Party: Principal Investigator, Miguel Sanchez Garcia, Director Critical Care, Hospital San Carlos, Madrid
Other Study IDs: Madrid COVID Tetrix
Record Dates: First submitted 2020-05-17; First posted 2020-05-19 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; ARDS, Human
Keywords: COVID-19; ARDS; Relocation; ICU capacity
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 9 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transferred patients: A subgroup of Critically ill intubated patients with COVID-19 associated ARDS were transferred from overwhelmed ICUs to other with available free beds
- Matched Non-transferred patients: A subgroup from the global cohort, matched for risk factors will be compared with transferred patients for outcome variables

SUMMARY:
Description of the adaptation of ICUs in the region of Madrid to que surge in demand of critical care due to COVID-19

DETAILED DESCRIPTION:
Background

The worldwide SARS-CoV-2 pandemic has put healthcare systems under the extreme pressure, with intensive care units being faced with a previously unseen number of patients with severe respiratory failure requiring admission for endotracheal intubation and mechanical ventilation.

Methods

The study describes how the critical care resources adapted to the sudden surge of severe Covid-19 in the province of Madrid, which developed at the beginning of March 2020. The response consisted of a swift increase in ICU capacity and the relocation of patients. ICU beds were mounted outside the usual intensive care areas. Transfer of critically ill intubated patients with COVID-19 was managed in an instant messenger service group composed of representatives of 53 intensive care units and performed by the Madrid Emergency Medical Systems (EMS). The investigators will compare transferred with non-transferred patients matched for risk factors for cardiovascular and respiratory complications.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to ICU in Madrid with COVID-19

Exclusion Criteria:

* Admitted to ICU without COVID-19

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill patients admitted to ICUs in Madrid for COVID-19
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2020-04-24 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | 9 weeks
  ICU mortality

SECONDARY OUTCOMES:
Length of ICU stay | 9 weeks
  From admission to discharge or death

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Sánchez García, MD, Principal Investigator — Hospital San Carlos, Madrid
Locations (1):
- Hospital Clinico San Carlos, Madrid, Spain